CLINICAL TRIAL: NCT07275606
Title: A Phase 1/2 Study of the Safety, Tolerability, and Pharmacokinetics of Cabotegravir in Neonates Exposed to HIV-1
Brief Title: A Study to Investigate Cabotegravir for Neonates Exposed to HIV-1
Acronym: CABNATE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 223560
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Cabotegravir; Neonate; HIV; Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a staggered design. There will be 2 stages with 2 cohorts in each. The 1st stage will focus on the oral CAB, the 2nd on the CAB LA injectable. In the 1st cohort at each stage, a single dose will be given. In the 2nd cohort of each stage, there will be a multi-dose regimen. Dose review decisions will be based upon safety, tolerability and pharmacokinetic data from each cohort.
Masking Description: Open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1: Single Oral Dose CAB (Cohort 1) group (Experimental): Participants receive a single dose of oral CAB suspension on study Day 1.
  Interventions: Drug: Oral CAB
- Stage 1: Multiple Oral Dose CAB (Cohort 2) group (Experimental): Participants receive repeat doses of oral CAB suspension starting on study Day 1. Dose and dosing frequency to be determined based on data from Cohort 1.
  Interventions: Drug: Oral CAB
- Stage 2: Single IM Dose CAB LA (Cohort 3) group (Experimental): Participants receive a single IM dose of CAB LA on study Day 1. Dose to be determined based on data from Cohort 2.
  Interventions: Drug: IM CAB LA
- Stage 2: Multiple IM Dose CAB LA (Cohort 4) group (Experimental): Participants receive repeat IM doses of CAB LA starting on study Day 1. Dose and dosing frequency to be determined based on data from Cohort 3.
  Interventions: Drug: IM CAB LA

INTERVENTIONS:
Drug: Oral CAB — CAB administered once orally on study Day 1 to the Stage 1: Single Oral Dose CAB (Cohort 1) and multiple times to the Stage 1: Multiple Oral Dose CAB (Cohort 2) group. Dose and dosing frequency for Cohort 2 to be determined based on emerging data from Cohort 1.
  Other Names: Cabotegravir
  Arms: Stage 1: Multiple Oral Dose CAB (Cohort 2) group; Stage 1: Single Oral Dose CAB (Cohort 1) group
Drug: IM CAB LA — CAB LA administered once intramuscularly on study Day 1 to the Stage 2: Single IM Dose CAB LA (Cohort 3) group and multiple times to the Stage 2: Multiple IM Dose CAB LA (Cohort 4) group, into the in the anterolateral thigh muscle of participants. Dose for Cohort 3 to be determined based on emerging data from Cohort 2. Dose and dosing frequency for Cohort 4 to be determined based on emerging data from Cohort 3.
  Other Names: Cabotegravir long-acting
  Arms: Stage 2: Multiple IM Dose CAB LA (Cohort 4) group; Stage 2: Single IM Dose CAB LA (Cohort 3) group

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of cabotegravir in neonates exposed to human immunodeficiency virus (HIV)-1.

ELIGIBILITY:
Inclusion Criteria:

* At least 37 weeks gestation at delivery.
* <=10 days of life.
* Birth weight at least 2 kg.
* At Entry, neonate has initiated standard of care Antiretroviral drug (ARV) prophylaxis.
* At Entry, neonate is generally healthy as determined by the site Investigator based on review of all available medical history information and physical examination findings.
* Mother is on a Dolutegravir (DTG) based regimen for a minimum of 4 weeks prior to delivery, regardless of maternal viral load.
* Mother is currently breastfeeding or plans to breastfeed infant.
* Mother is of legal age or circumstance to provide independent informed consent and is willing and able to provide documented informed consent for her and her infant's participation in this study.
* Mother has confirmed HIV-1 infection based on positive test results from 2 samples collected from 2 separate blood samples. Test results may be obtained from medical records or from testing performed during the study Screening period.

Exclusion Criteria:

Medical conditions

* Severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by examining clinician.
* Known maternal-fetal blood group incompatibility which can result in hemolytic disease of the newborn.
* Known family history of G6PD deficiency.
* Prior/Concomitant therapy
* Mother who has previously received, is receiving, or will be receiving CAB post-partum.
* Neonate or breastfeeding mother is receiving any disallowed medication.
* Prior/Concurrent clinical study participation
* Neonate has exposure to other investigational drugs that might interfere with study intervention metabolism.
* Diagnostic assessments
* Mother has known Integrase strand transfer inhibitor (InSTI) resistance.
* At Entry, neonate with a confirmed, documented positive HIV Nucleic acid amplification test (NAAT) test result.
* At Screening, neonate has any of the following laboratory test results:

  * Alanine transaminase or Aspartate aminotransferase of more than 2.5 x Upper limit of normal (ULN).
  * Total bilirubin in range for phototherapy at Entry.
  * Hemoglobin <13.0 g/dL.
  * Decreased white blood cells Grade 3 or above.
  * Platelets <50 000 cells/mm3
  * Creatinine value more than 1.3 the ULN for postnatal age as defined in Division of AIDS (DAIDS)
  * Albumin Grade 3 or higher.
  * Direct bilirubin Grade 3 and above.
* Any other Grade ≥3 event on DAIDS toxicity table
* Neonates with prior exchange transfusion. Other exclusion criteria
* Mother or neonate has a condition that, in the site Investigator or designee's opinion, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Neonate is receiving DTG as part of HIV prophylactic regimen. Liver safety exclusion criteria
* Known maternal hepatitis B infection. Cardiac safety exclusion criteria
* At screening, QT interval corrected using Fridericia's formula >450 msec.

Max Age: 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2026-03-17 (Estimated); Primary Completion 2029-10-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of CAB in participants from Stage 1: Single Oral Dose CAB (Cohort 1) group | At study Days 1, 3, 8, 15 and 22
  Blood samples are collected at specific time points for PK analysis to determine Cmax.
Maximum observed plasma concentration (Cmax) of CAB LA in participants from Stage 2: Single IM Dose CAB LA (Cohort 3) group | At study Days 1, 3, 9,16, 28 and 42
  Blood samples are collected at specific time points for PK analysis to determine Cmax.
Last observed plasma concentration (Clast) of CAB in participants from Stage 1: Single Oral Dose CAB (Cohort 1) group | At study Days 1, 3, 8, 15 and 22
  Blood samples are collected at specific time points for PK analysis to determine Clast.
Last observed plasma concentration (Clast) of CAB LA in participants from Stage 2: Single IM Dose CAB LA (Cohort 3) group | At study Days 1, 3, 9, 16, 28 and 42
  Blood samples are collected at specific time points for PK analysis to determine Clast.
Area under the curve time 0 to the last time point (AUC0-t) of CAB in participants from Stage 1: Single Oral Dose CAB (Cohort 1) group | At study Days 1, 3, 8, 15 and 22
  Blood samples are collected at specific time points for PK analysis to determine AUC0-t.
Area under the curve time 0 to the last time point (AUC0-t) of CAB LA in participants from Stage 2: Single IM Dose CAB LA (Cohort 3) group | At study Days 1, 3, 9, 16, 28 and 42
  Blood samples are collected at specific time points for PK analysis to determine AUC0-t.
Pre-dose concentrations (C0h) of CAB in participants from Stage 1: Multiple Oral Dose CAB (Cohort 2) group | At Study Days 1, 3, 7, 14, 28, 35, 42 and 49
  Blood samples are collected at specific time points for PK analysis to determine C0h.
Pre-dose concentrations (C0h) of CAB LA in participants from Stage 2: Multiple IM Dose CAB LA (Cohort 4) group | At Study Days 1, 3, 7, 21, 28, 42, 56, 70, 84, 98, 112, 140 and 168
  Blood samples are collected at specific time points for PK analysis to determine C0h.
Post-dose concentrations of CAB in participants from Stage 1: Multiple Oral Dose CAB (Cohort 2) group | At Study Days 1, 3, 7, 14, 21, 28, 35, 42 and 49
  Blood samples are collected at specific time points for PK analysis to determine post-dose concentrations.
Post-dose concentrations of CAB LA in participants from Stage 2: Multiple IM Dose CAB LA (Cohort 4) group | At Study Days 1, 3, 7, 14, 21, 28, 35, 42, 56, 70, 84, 98, 112, 140 and 168
  Blood samples are collected at specific time points for PK analysis to determine post-dose concentrations.
Number of participants with drug-related adverse event (AEs) by severity | From Day 1 up to 2-months post last dose administration (last dose administered at Day 1 to the single dose groups, at Month 1 to Stage 1: Multiple Oral Dose CAB (Cohort 2) group and at Month 6 to Stage 2: Multiple IM Dose CAB LA (Cohort 4) group)
  A drug-related AE is any untoward medical occurrence in a clinical study participant considered related to the study intervention. The severity of events is graded using the DAIDS grading scale, where grades are defined based on numeric criteria as follows: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life-threatening. A higher grade indicates greater severity.
Number of participants with serious AEs (SAEs) by severity | From Day 1 up to 2-months post last dose administration (last dose administered at Day 1 to the single dose groups, at Month 1 to Stage 1: Multiple Oral Dose CAB (Cohort 2) group and at Month 6 to Stage 2: Multiple IM Dose CAB LA (Cohort 4) group)
  An SAE is defined as any untoward medical occurrence that is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in death.
  The severity of events is graded using the DAIDS grading scale, where grades are defined based on numeric criteria as follows: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life-threatening. A higher grade indicates greater severity.
Number of participants with injection site reactions (ISRs) by severity | From Day 1 up to 2-months post last dose administration (last dose administered at Day 1 to the single dose groups, at Month 1 to Stage 1: Multiple Oral Dose CAB (Cohort 2) group and at Month 6 to Stage 2: Multiple IM Dose CAB LA (Cohort 4) group)
  An ISR is defined as an adverse event which is localized at the injection site, typically includes pain, tenderness, erythema, redness, induration, swelling, nodules or pruritus, but may also encompass other reactions. The severity of events is graded using the DAIDS grading scale, where grades are defined based on numeric criteria as follows: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life-threatening. A higher grade indicates greater severity.
Number of participants who discontinue the study intervention due to AEs or injection intolerability | From Day 1 up to 2-months post last dose administration (last dose administered at Day 1 to the single dose groups, at Month 1 to Stage 1: Multiple Oral Dose CAB (Cohort 2) group and at Month 6 to Stage 2: Multiple IM Dose CAB LA (Cohort 4) group)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Number of participants developing Grade 3 and higher AEs and SAEs, by severity | From Day 1 up to 2-months post last dose administration (last dose administered at Day 1 to the single dose groups, at Month 1 to Stage 1: Multiple Oral Dose CAB (Cohort 2) group and at Month 6 to Stage 2: Multiple IM Dose CAB LA (Cohort 4) group)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in death. The severity of events is graded using the DAIDS grading scale, where grades are defined based on numeric criteria as follows: Grade 3 = severe and Grade 4 = potentially life-threatening. A higher grade indicates greater severity.
Number of participants with Grade 3 and above bilirubin elevation. | From Day 1 up to 2-months post last dose administration (last dose administered at Day 1 to the single dose groups, at Month 1 to Stage 1: Multiple Oral Dose CAB (Cohort 2) group and at Month 6 to Stage 2: Multiple IM Dose CAB LA (Cohort 4) group)
  The severity of events is graded using the DAIDS grading scale, where grades are defined based on numeric criteria as follows: Grade 3 = severe and Grade 4 = potentially life-threatening. A higher grade indicates greater severity.

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf